CLINICAL TRIAL: NCT01915511
Title: Idiopathic Pulmonary Fibrosis Prospective Outcomes (IPF-PRO) and Interstitial Lung Disease Prospective Outcomes (IPF-PRO/ILD-PRO) Registry
Brief Title: Idiopathic Pulmonary Fibrosis and Interstitial Lung Disease Prospective Outcomes Registry
Acronym: IPF/ILD-PRO
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00046131; 1199.174 (Other: DCRI)
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis, Interstitial Lung Disease
Keywords: Idiopathic pulmonary fibrosis; Pulmonary fibrosis; IPF; Registry; 1199.174; Interstitial Lung Disease; ILD; Interstitial Lung Disease with Progressive Phenotype
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood for DNA collected at enrollment. Plasma, serum, and RNA samples collected at enrollment and approximate 6-month intervals throughout study follow-up.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subjects with a new IPF diagnosis: Subjects with a new diagnosis of IPF established at the time of enrollment in the registry
- Subjects with a non-IPF ILD diagnosis: Subjects with a diagnosis of a non-IPF ILD of any duration, including, but not limited to Idiopathic Non-Specific Interstitial Pneumonia (iNSIP), Unclassifiable Idiopathic Interstitial Pneumonias (IIPs), Interstitial Pneumonia with Autoimmune Features (IPAF), Autoimmune ILDs such as Rheumatoid Arthritis (RA-ILD) and Systemic Sclerosis (SSc-ILD), Chronic Hypersensitivity Pneumonitis (HP), Sarcoidosis or Exposure-related ILDs such as asbestosis with progressive phenotype
- New Subjects with a new IPF diagnosis: Subjects with a new diagnosis of IPF established at the time of enrollment in the registry not previously enrolled in the registry.

SUMMARY:
The Idiopathic Pulmonary Fibrosis Prospective Outcomes (IPF-PRO) Registry started recruiting in 2014 with the objective of studying Idiopathic Pulmonary Fibrosis. In 2018, the registry expanded to include recruitment of participants with other chronic fibrosing interstitial lung diseases (ILDs) with progressive phenotype also referred to as progressive fibrosing interstitial lung diseases in the Chronic Fibrosis Interstitial Lung Disease with Progressive Phenotype (ILD-PRO) Registry. When the third phase of the registry begins, the IPF-PRO registry will enroll additional patients with idiopathic pulmonary fibrosis. This IPF-PRO registry is a prospective registry that will collect information regarding the natural history, health care interactions, participant reported questionnaire data to assess quality of life, and the methods of treatment of participants with a diagnosis of idiopathic pulmonary fibrosis (IPF) or of another chronic fibrosing interstitial lung disease (ILD) with progressive phenotype established at the enrolling centers. In addition, blood samples and chest image studies will be collected and banked for future research projects.

DETAILED DESCRIPTION:
This registry originally enrolled a total of 1002 participants newly diagnosed with IPF and continues to enroll patients with other chronic fibrosing ILDs with newly identified progressive phenotype to reach an enrollment of 1000 patients. Participants will be enrolled in three phases, (IPF-PRO and ILD-PRO) over a span of 8 years at approximately 50 sites experienced in the diagnosis and treatment of ILD in the United States. Enrollment for the original IPF cohort started in 2014 and ended in October 2018, with 1002 total participants enrolled. In the third phase of the registry new enrollment for patients with IPF will restart in 2023-2024 with the plan to enroll up to 1000 new IPF patients, for a total IPF enrollment of 2000. Enrollment for other chronic fibrosing ILDs with newly identified progressive phenotype cohort was initiated in February 2019 and will end when enrollment reaches 1000 participants with the potential of enrolling another 1000 participants with other chronic fibrosing ILDs with newly identified without a progressive phenotype. Data and samples will be collected from participants for approximately 5 years for the IPF cohort. For the chronic fibrosing ILD with progressive phenotype cohort, data and samples will be collected for a minimum of 3 years, up to approximately 5 years. Participant management and treatment decisions will be determined by participants and their health care professionals.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Established a new diagnosis (within 12 months) of IPF by the enrolling center.
* Age 21 years or older, or
* Diagnosis of a non-IPF ILD of any duration, including, but not limited to Idiopathic Non-Specific Interstitial Pneumonia (iNSIP), Unclassifiable Idiopathic Interstitial Pneumonias (IIPs), Interstitial Pneumonia with Autoimmune Features (IPAF), Autoimmune ILDs such as Rheumatoid Arthritis (RA-ILD) and Systemic Sclerosis (SSc-ILD), Chronic Hypersensitivity Pneumonitis (HP), Sarcoidosis or Exposure-related ILDs such as asbestosis with progressive phenotype during the last 24 months by the enrolling center that meets the following criteria:

  * Chronic fibrosing ILD as defined by reticular abnormality with traction bronchiectasis with or without honeycombing confirmed by chest HRCT scan and/or lung biopsy.
  * Progressive phenotype as defined by fulfilling at least one of the criteria below of fibrotic changes (progression set point) within the last 24 months regardless of treatment considered appropriate in individual ILDs (8):

    * decline in FVC % predicted (% pred) based on ≥10% relative decline
    * decline in FVC % pred based on ≥5 - <10% relative decline in FVC combined with worsening of respiratory symptoms as assessed by the site investigator
    * decline in FVC % pred based on ≥5 - <10% relative decline in FVC combined with increasing extent of fibrotic changes on chest imaging (HRCT scan) as assessed by the site investigator
    * decline in DLCO % pred based on≥ 10% relative decline
    * worsening of respiratory symptoms as well as increasing extent of fibrotic changes on chest imaging (HRCT scan) as assessed by the site investigator independent of FVC change.

The relative decline for FVC % predicted is calculated using the formula:

Relative Decline= (FVC % Pred (Reference)-FVC % Pred (Screening))/(FVC % Pred (Reference))×100%, where FVC % Pred (Reference) is the greatest measurement of FVC % predicted in the 24 months prior to screening and FVC % Pred (Screening) is the measurement of FVC % predicted at screening.

The relative decline for DLCO % predicted is calculated using the formula:

Relative Decline= (DLCO % Pred (Reference)-DLCO % Pred (Screening))/(DLCO % Pred (Reference))×100%, Where DLCO % Pred (Reference) is the greatest measurement of DLCO % Pred in the 24 months prior to screening and DLCO % Pred (Screening) is the measurement of DLCO % Pred at screening

Exclusion Criteria:

* Malignancy, treated or untreated, other than skin or early -stage prostate cancer, within the past 5 years
* Currently listed for lung transplantation at the time of enrollment
* Currently enrolled in an interventional clinical trial at the time of enrollment in this registry
* For the additional IPF cohort of 1000 individuals, previous enrollment in this registry.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a new diagnosis of IPF or a non- IPF chronic fibrosing ILD established at the time of enrollment in the registry are eligible for participation in the IPF-PRO/ILD-PRO registry if the participant meets the selection criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-06; Primary Completion 2028-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Data on natural history of IPF & non-IPF chronic fibrosing ILD | End of Study (3 years after last patient will be enrolled)
  Characterize and describe the natural history of patients with a recent confirmed diagnosis of IPF, with emphasis on demographics, co-morbidities, medications, and risks for disease progression or death.
Data on current practice patterns for diagnosis of IPF & non-IPF chronic fibrosing ILD | End of Study (3 years after last patient will be enrolled)
  Understand the current practice patterns for diagnosis of IPF & non-IPF chronic fibrosing ILD
Data on impact of IPF & non- IPF chronic fibrosing ILD on patient quality of life. | End of Study (3 years after last patient will be enrolled)
  Describe the impact of IPF & non- IPF chronic fibrosing ILD on patient quality-of-life (QOL).
Blood samples for future research. | End of Study (3 years after last patient will be enrolled)
  Collect longitudinal bio-samples for future research on disease presentation, progression, and subject response to clinical interventions.
HRCT images for future research (for non-IPF chronic fibrosing ILD, and new IPF patients cohort) | End of Study (3 years after last patient will be enrolled)
  Collect longitudinal HRCT images for future research

SECONDARY OUTCOMES:
Data on management practices compared to existing guidelines. | End of Study (3 years after last patient will be enrolled)
  Compare disease-specific management practices with existing guidelines.
Data on center-specific practices on outcomes. | End of Study (3 years after last patient will be enrolled)
  Determine the influence of center-specific practices on patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Palmer, MD, Principal Investigator — Duke Clinical Research Institute, Duke University
Locations (41):
- United States (41):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of California - Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Healthcare, Austell, Georgia
  - University of Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Loyola University Health System, Maywood, Illinois
  - University of Kansas, Kansas City, Kansas
  - Tulane University, New Orleans, Louisiana
  - University from Virginia, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - NYU Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Pulmonix LLC, Greensboro, North Carolina
  - PMG Research, Wilmington, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Clinic, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Baylor University Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Lung Center, Houston, Texas
  - Inova, Falls Church, Virginia
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Menon AA, Gansen B, Mulder H, Neely ML, Papavasileiou P, Salisbury ML, Southern BD, Hesslinger C, Leonard TB, Meissner F, Todd JL. Mass spectrometry-based peripheral blood proteomics for biomarker discovery in idiopathic pulmonary fibrosis. Respir Res. 2025 Oct 22;26(1):294. doi: 10.1186/s12931-025-03377-5. PMID 41126189
- [Derived] Swaminathan AC, Weber JM, Todd JL, Palmer SM, Neely ML, Whelan TP, Kim GHJ, Leonard TB, Goldin J. Extent of lung fibrosis is of greater prognostic importance than HRCT pattern in patients with progressive pulmonary fibrosis: data from the ILD-PRO registry. Respir Res. 2025 Feb 28;26(1):73. doi: 10.1186/s12931-025-03136-6. PMID 40022059
- [Derived] Oldham JM, Neely ML, Wojdyla DM, Gulati M, Li P, Patel DC, Palmer SM, Todd JL; IPF-PRO Registry Investigators. Changes in Lung Function and Mortality Risk in Patients With Idiopathic Pulmonary Fibrosis. Chest. 2025 Aug;168(2):415-422. doi: 10.1016/j.chest.2025.02.018. Epub 2025 Feb 26. PMID 40020995
- [Derived] Sack C, Wojdyla DM, MacMurdo MG, Gassett A, Kaufman JD, Raghu G, Redlich CA, Li P, Olson AL, Leonard TB, Todd JL, Neely ML, Snyder LD, Gulati M; IPF-PRO Registry investigators. Long-Term Air Pollution Exposure and Severity of Idiopathic Pulmonary Fibrosis: Data from the Idiopathic Pulmonary Fibrosis Prospective Outcomes (IPF-PRO) Registry. Ann Am Thorac Soc. 2025 Mar;22(3):378-386. doi: 10.1513/AnnalsATS.202404-382OC. PMID 39531618
- [Derived] Wang L, Wu P, Liu Y, Patel DC, Leonard TB, Zhao H. Clustering-aided prediction of outcomes in patients with idiopathic pulmonary fibrosis. Respir Res. 2024 Oct 23;25(1):383. doi: 10.1186/s12931-024-03015-6. PMID 39443991
- [Derived] Lobo LJ, Liu Y, Li P, Ramaswamy M, Swaminathan AC, Veeraraghavan S, Fan Y, Neely ML, Palmer SM, Olson AL; ILD-PRO Registry investigatorsdagger. Design and baseline characteristics of the ILD-PRO registry in patients with progressive pulmonary fibrosis. BMC Pulm Med. 2024 Sep 27;24(1):468. doi: 10.1186/s12890-024-03247-8. PMID 39334205
- [Derived] Summer R, Todd JL, Neely ML, Lobo LJ, Namen A, Newby LK, Shafazand S, Suliman S, Hesslinger C, Keller S, Leonard TB, Palmer SM, Ilkayeva O, Muehlbauer MJ, Newgard CB, Roman J. Circulating metabolic profile in idiopathic pulmonary fibrosis: data from the IPF-PRO Registry. Respir Res. 2024 Jan 25;25(1):58. doi: 10.1186/s12931-023-02644-7. PMID 38273290
- [Derived] Neely ML, Hellkamp AS, Bender S, Todd JL, Liesching T, Luckhardt TR, Oldham JM, Raj R, White ES, Palmer SM. Lung function trajectories in patients with idiopathic pulmonary fibrosis. Respir Res. 2023 Aug 24;24(1):209. doi: 10.1186/s12931-023-02503-5. PMID 37612608
- [Derived] Ruan P, Todd JL, Zhao H, Liu Y, Vinisko R, Soellner JF, Schmid R, Kaner RJ, Luckhardt TR, Neely ML, Noth I, Porteous M, Raj R, Safdar Z, Strek ME, Hesslinger C, Palmer SM, Leonard TB, Salisbury ML. Integrative multi-omics analysis reveals novel idiopathic pulmonary fibrosis endotypes associated with disease progression. Respir Res. 2023 May 31;24(1):141. doi: 10.1186/s12931-023-02435-0. PMID 37344825
- [Derived] Swaminathan AC, Hellkamp AS, Neely ML, Bender S, Paoletti L, White ES, Palmer SM, Whelan TPM, Dilling DF; Idiopathic Pulmonary Fibrosis Prospective Outcomes Registry investigators. Disparities in Lung Transplant among Patients with Idiopathic Pulmonary Fibrosis: An Analysis of the IPF-PRO Registry. Ann Am Thorac Soc. 2022 Jun;19(6):981-990. doi: 10.1513/AnnalsATS.202105-589OC. PMID 35073248
- [Derived] Kim HJ, Snyder LD, Neely ML, Hellkamp AS, Hotchkin DL, Morrison LD, Bender S, Leonard TB, Culver DA; IPF-PRO Registry investigators. Clinical Outcomes of Patients with Combined Idiopathic Pulmonary Fibrosis and Emphysema in the IPF-PRO Registry. Lung. 2022 Feb;200(1):21-29. doi: 10.1007/s00408-021-00506-x. Epub 2022 Jan 7. PMID 34997268
- [Derived] de Andrade JA, Kulkarni T, Neely ML, Hellkamp AS, Case AH, Culver DA, Guntupalli K, Bender S, Conoscenti CS, Snyder LD; IPF-PRO Registry Investigators. Associations between resources and practices of ILD centers and outcomes in patients with idiopathic pulmonary fibrosis: data from the IPF-PRO Registry. Respir Res. 2022 Jan 7;23(1):3. doi: 10.1186/s12931-021-01921-7. PMID 34996465
- [Derived] Kim HJ, Snyder LD, Adegunsoye A, Neely ML, Bender S, White ES, Conoscenti CS, Strek ME; IPF-PRO Registry Investigators. Hospitalizations in patients with idiopathic pulmonary fibrosis. Respir Res. 2021 Sep 30;22(1):257. doi: 10.1186/s12931-021-01851-4. PMID 34592998
- [Derived] Salisbury ML, Conoscenti CS, Culver DA, Yow E, Neely ML, Bender S, Hartmann N, Palmer SM, Leonard TB; IPF-PRO Registry principal investigators as follows. Antifibrotic Drug Use in Patients with Idiopathic Pulmonary Fibrosis. Data from the IPF-PRO Registry. Ann Am Thorac Soc. 2020 Nov;17(11):1413-1423. doi: 10.1513/AnnalsATS.201912-880OC. PMID 32574517
- [Derived] Fan Y, Bender SD, Conoscenti CS, Davidson-Ray L, Cowper PA, Palmer SM, de Andrade JA; IPF-PRO Registry Investigators. Hospital-Based Resource Use and Costs Among Patients With Idiopathic Pulmonary Fibrosis Enrolled in the Idiopathic Pulmonary Fibrosis Prospective Outcomes (IPF-PRO) Registry. Chest. 2020 Jun;157(6):1522-1530. doi: 10.1016/j.chest.2019.12.041. Epub 2020 Jan 29. PMID 32004554
- [Derived] O'Brien EC, Hellkamp AS, Neely ML, Swaminathan A, Bender S, Snyder LD, Culver DA, Conoscenti CS, Todd JL, Palmer SM, Leonard TB; IPF-PRO Registry investigators. Disease Severity and Quality of Life in Patients With Idiopathic Pulmonary Fibrosis: A Cross-Sectional Analysis of the IPF-PRO Registry. Chest. 2020 May;157(5):1188-1198. doi: 10.1016/j.chest.2019.11.042. Epub 2020 Jan 15. PMID 31954102
- [Derived] Todd JL, Neely ML, Overton R, Durham K, Gulati M, Huang H, Roman J, Newby LK, Flaherty KR, Vinisko R, Liu Y, Roy J, Schmid R, Strobel B, Hesslinger C, Leonard TB, Noth I, Belperio JA, Palmer SM; IPF-PRO Registry investigators. Peripheral blood proteomic profiling of idiopathic pulmonary fibrosis biomarkers in the multicentre IPF-PRO Registry. Respir Res. 2019 Oct 22;20(1):227. doi: 10.1186/s12931-019-1190-z. PMID 31640794
- [Derived] Snyder L, Neely ML, Hellkamp AS, O'Brien E, de Andrade J, Conoscenti CS, Leonard T, Bender S, Gulati M, Culver DA, Kaner RJ, Palmer S, Kim HJ; IPF-PRO Registry investigators. Predictors of death or lung transplant after a diagnosis of idiopathic pulmonary fibrosis: insights from the IPF-PRO Registry. Respir Res. 2019 May 30;20(1):105. doi: 10.1186/s12931-019-1043-9. PMID 31142314
- [Derived] O'Brien EC, Durheim MT, Gamerman V, Garfinkel S, Anstrom KJ, Palmer SM, Conoscenti CS. Rationale for and design of the Idiopathic Pulmonary Fibrosis-PRospective Outcomes (IPF-PRO) registry. BMJ Open Respir Res. 2016 Jan 11;3(1):e000108. doi: 10.1136/bmjresp-2015-000108. eCollection 2016. PMID 26835134